CLINICAL TRIAL: NCT00036543
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study of the Safety and Efficacy of 10 Mg Atrasentan in Men With Metastatic, Hormone-Refractory Prostate Cancer
Brief Title: A Study of Atrasentan in Men With Metastatic, Hormone-Refractory Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M00-211; NCT00026481 (obsolete NCT alias)
Record Dates: First submitted 2002-05-10; First posted 2002-05-13 (Estimated); Last update posted 2006-08-15 (Estimated); Status verified 2006-08

CONDITIONS: Prostate Cancer
Keywords: Hormone-Refractory, Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Atrasentan

INTERVENTIONS:
Drug: Atrasentan

SUMMARY:
This study is being done to evaluate the safety and efficacy of atrasentan in men with metastatic hormone-refractory prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of prostate cancer.
* Rising PSA while on hormonal therapy or following surgical castration.
* Documented evidence of metastatic disease.

Exclusion Criteria:

* Have received cytotoxic chemotherapy.
* Have received opioid or narcotic medications (such as codeine or morphine) or radiation for pain caused by your prostate cancer in the last 6 months.

Min Age: 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000
Dates: Start 2001-05

PRIMARY OUTCOMES:
The primary objective of this study is to evaluate safety and efficacy as measured by time-to-disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Darryl Sleep, M.D., Study Director — Abbott
Locations (232):
- United States (79):
  - Urology Centers Of Alabama, Homewood, Alabama
  - Alaska Clinical Research Center, LLC, Anchorage, Alaska
  - Advanced Clinical Trials, Tucson, Arizona
  - Arkansas Urologial Associates, PA, Little Rock, Arkansas
  - Robin V. Smith, MD, Chula Vista, California
  - Urology Associate Of Central California, Fresno, California
  - South Valley Medical Plaza, Gilroy, California
  - San Diego Urology Center, La Mesa, California
  - UCLA School Of Medicine, Los Angeles, California
  - Hillcrest Urological Medical Group, Inc., San Diego, California
  - Urology Associates Of San Luis Obispo, San Luis Obispo, California
  - Pacific Clinical Research, Santa Monica, California
  - Western Clinical Research, Inc., Torrance, California
  - Urology Associate, Pc, Denver, Colorado
  - South Fl Medical Research, Aventura, Florida
  - Clinical Physiology Associates, Fort Myers, Florida
  - Advanced Research Institute, New Port Richey, Florida
  - Urology Treatment Center, Sarasota, Florida
  - Southeastern Urological Center, P.A., Tallahassee, Florida
  - Winship Cancer Institute Emory University, Atlanta, Georgia
  - Sandy Springs Urology, Atlanta, Georgia
  - Atlanta Va Medical Center, Decatur, Georgia
  - Dreyer Medical Clinic, Aurora, Illinois
  - Progressive Care, S.C., Chicago, Illinois
  - Weiss Memorial Hospital, Chicago, Illinois
  - Evanston Hospital Kellogg Cancer Center, Evanston, Illinois
  - Welborn Clinic, Evansville, Indiana
  - Urologic Associates, Pc, Davenport, Iowa
  - Iowa Urology, Des Moines, Iowa
  - Kansas University Medical Center, Kansas City, Kansas
  - Ochsner Clinic, Department of Urology, New Orleans, Louisiana
  - Regional Urology, Shreveport, Louisiana
  - LSUHSC, Shreveport, Louisiana
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - Mid Atlantic Clinical Research, Rockville, Maryland
  - Michigan Institute Of Urology, Pc, Saint Clair Shores, Michigan
  - Lakeside Urology, PC, Saint Joseph, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - The Medical Oncology Group, Gulfport, Mississippi
  - St. Joseph Oncology, Saint Joseph, Missouri
  - Washington University, St Louis, Missouri
  - Billings Oncology Associates, Billings, Montana
  - Nevada Urology Associate, Reno, Nevada
  - Albany Medical Center South Clinical Campus, Albany, New York
  - HemOnCare, PC, Brooklyn, New York
  - Beth Israel Medical Center, New York, New York
  - NYU Medical Center, New York, New York
  - Nyack Hospital, Nyack, New York
  - Rochester General Hospital, Rochester, New York
  - St. Vincent's Medical Center - Staten Island, Staten Island, New York
  - Albert Einstein College of Medicine, The Bronx, New York
  - The University Of North Carolina At Chapel Hill, Chapel Hill, North Carolina
  - Blumenthal Cancer Center, Charlotte, North Carolina
  - The Urology Center, Greensboro, North Carolina
  - Urologic Specialists Of Oklahoma, Inc., Tulsa, Oklahoma
  - Oregon Urology Specialists, Eugene, Oregon
  - Urologic Associates of Allentown, Allentown, Pennsylvania
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Urological Associates Of Lancaster, Lancaster, Pennsylvania
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - University Of Pittsburgh, Pittsburgh, Pennsylvania
  - Center for Urologic Care, West Reading, Pennsylvania
  - Urology Associates, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Dept of Veteran's Affairs North Texas Healthcare System, Dallas, Texas
  - Ntouch Research Corporation, Dallas, Texas
  - Uthscsa, San Antonio, Texas
  - Scott & White Memorial Hospital, Temple, Texas
  - Anthony Middleton, M.D., Salt Lake City, Utah
  - Western Urological Clinic, Salt Lake City, Utah
  - University Of Vermont, Burlington, Vermont
  - Virginia Urology Center, Richmond, Virginia
  - Seattle Urological Associates, Seattle, Washington
  - University Of Washington School Of Medicine, Seattle, Washington
  - Jeffrey Frankel, M.D., Seattle, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - Midwest Research Specialists, LLC, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Wyoming Research Foundation, Cheyenne, Wyoming
- Australia (10):
  - St Vincent's Clinic, Darlinghurst, New South Wales
  - Prince Of Wales Hospital, Randwick, New South Wales
  - Westmead Public Hospital, Westmead, New South Wales
  - Royal Brisbane Hospital, Herston, Queensland
  - Repatriation General Hospital, Daws Park, South Australia
  - Peter Maccallum Cancer Institute, East Melbourne, Victoria
  - Bayside Urology, Mentone, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Hollywood Specialist Centre, Nedlands, Western Australia
  - Princess Alexandra Hospital, Woolloongabba
- Austria (3):
  - Universitatsklinik Innsbruck, Innsbruck
  - Urologische Abteilung, Linz
  - Landesklinik fur Urologie und Andrologie, Salzburg
- Belgium (8):
  - A.Z. Middelheim, Antwerp
  - AZ Middelheim, Antwerp
  - A Z St Jan, Bruges
  - University Hospital Erasme, Brussels
  - Uz Gent, Ghent
  - Virga Jesse Hospital, Hasselt
  - C.H.U. Liege, Liège
  - St-Elisabeth Ziekenhuis, Turnhout
- Canada (26):
  - Tom Baker Cancer Center, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Wilson Urology, Kelowna, British Columbia
  - Dr. Cal Andreou, Surrey, British Columbia
  - Vancouver Hospital & Health Sciences Centre, Vancouver, British Columbia
  - Dr. P. J. Pommerville, Inc., Victoria, British Columbia
  - Dr. Gary Steinhoff, Clinical Research, Victoria, British Columbia
  - Abbott Clinic, Winnipeg, Manitoba
  - Queen Elizabeth II Health Sciences Center, Halifax, Nova Scotia
  - Valley Professional Centre, Kentville, Nova Scotia
  - The Male Health Centres, Barrie, Ontario
  - Burlington Professional Centre, Burlington, Ontario
  - The Urology Resource Centre, Burlington, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - Probidity Medical Research, Kitchener, Ontario
  - London Health Sciences Centre, London, Ontario
  - Quest Clinical Trials, Markham, Ontario
  - Walk-In Clinic, North Bay, Ontario
  - Jack Barkin, M.D., North York, Ontario
  - The Male Health Centres, Oakville, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Service Radio-Oncologie, Chus, Fleurimont, Quebec
  - Hopital Notre-Dame, Montreal, Quebec
  - Royal Victoria Hospital, Montreal, Quebec
  - Ultramed, Pointe-Claire, Quebec
  - Chuq Pavillon Hotel-Dieu, Québec, Quebec
- France (7):
  - Hopital De Pontchaillou, Rennes, Cedex
  - Hopital De Rangueil, Toulouse, Cedex
  - CHU Hôpital Côte De Nacre, Caen
  - Hôpital Henri Mondor, Créteil
  - CHU de Bicêtre, Le Kremlin-Bicêtre
  - Hopital Bichat Claude Bernard, Paris
  - Hôpital Foch, Suresnes
- Germany (15):
  - Krankenhaus Am Urban, Berlin
  - Allgemeines Krankenhaus Urologie, Celle
  - Universitätsklinikum Carl Gustav Carus an der, Dresden
  - Universitätsklinikum Urologie, Essen
  - Universitätsklinkum, Freiburg im Breisgau
  - Allgemeines Krankenhaus Barmbek, Hamburg
  - Klinik Und Poliklinik für Urologie und Kinder, Homburg / SAAR
  - Universitutsklinikum Lubeck Urologie, Lübeck
  - Universitätsklinikum Mannheim, Mannheim
  - Urologische Klinik Und Poliklinik Grosshadern, München
  - Klinikum Rechts Der Isar, München
  - Universitätsklinikum, Münster
  - Städtische Kliniken, Urologie, Offenbach
  - Universitat Ulm, Ulm
  - Klinikum Wuppertal GmbH, Wuppertal
- Greece (3):
  - 'Alexandra' Hospital, Athens
  - Pe.Pa.G.N.I Hospital, Heraklion
  - G. Genimatas Hospital, Thessaloniki
- Ireland (3):
  - Tallaght Hospital, Dublin
  - St Vincent'S Hospital, Dublin
  - Mater Misericordiae Hospital, Dublin
- Italy (6):
  - Clinica Urologica I - Università di Bari, Bari
  - Istituto Nazionale per la Ricerca sul Cancro -IST, Genoa
  - Istituto Europeo di Oncologia, Milan
  - Clinica Urologica - Università Di Milano, Milan
  - Istituto di Urologia, Padua
  - Policlinico G. B. Rossi, Verona
- Netherlands (8):
  - Amc, Amsterdam
  - Rijnstate Hospital, Arnhem
  - Medisch Spectrun Twente, Enschede
  - Atrium Heerlen, Heerlen
  - University Hospital Maastricht, Maastricht
  - University Hospital Rotterdam, Rotterdam
  - St Franciscus Gasthuis, Rotterdam
  - University Hospital Utrecht, Utrecht
- New Zealand (2):
  - Canterbury Urology Research Trust, Christchurch
  - Promed Urology Ltd., Tauranga
- Poland (5):
  - Katedra I Klinika Urologi AM, Gdansk
  - Katedra i Klinika Urologii - Akademia Medyczna w Gdansku, Gdansk
  - Samodzielny Publiczny Zaklad Opieki, Katowice
  - Szpital Kliniczny Dzieciatka Jezus, Warsaw
  - Akademia Medyczna we Wroclawiu, Wroclaw
- South Africa (9):
  - Mediclinic Hospital, Petermaritzburg, 3201
  - Constantiaberg Medi-Clinic, Cape Town
  - University Of Stellenbosch, Cape Town
  - University Of Natal - Nelson R Mandela School of Medicine, Durban
  - Kenridge St Joseph Wingl, Parktown
  - Medi-Clinic Hospital, Pietermaritzburg
  - Medical Centre, Pietermaritzburg
  - Pretoria Urology Hospital, Pretoria
  - Pretoria Academic Hospital, Pretoria
- Spain (10):
  - Hospital Juan Canalejo, A Coruña
  - Fundacion Puigvert, Barcelona
  - Hospital Vall D'Hebron, Barcelona
  - Hospital de Galdakao, Galdakao-Vizcaya
  - Hospital Gregorio Maranon, Madrid
  - Clinica Puerta De Hierro, Madrid
  - Hospital 12 De Octubre, Madrid
  - Hospital Carlos Haya, Málaga
  - Hospital Marques De Valdecilla, Santander
  - Instituto Valenciano De Oncologia, Valencia
- Sweden (9):
  - Sahlgrenska University Hospital, Gothenburg
  - Helsingborg Hospital, Helsingborg
  - Linkoping University Hospital, Linköping
  - Lund University Hospital, Lund
  - Malmo University Hospital MAS, Malmo
  - Orebro Regional Hospital, Örebro
  - Karolinska Hospital, Stockholm
  - Umea University Hospital, Umeå
  - Uppsala University Hospital, Uppsala
- Switzerland (3):
  - Zentrum fur Onkologie, Hämatologie und, Aarau
  - Inselspital, Universität Bern, Bern
  - Chefarzt Urologische Klinik - Universitätsspital Zürich, Zurich
- United Kingdom (26):
  - Royal Devon And Exeter Hospital, Exeter, Devon
  - Lister Hospital, Stevenage, Hertfordshire
  - Northwick Park Hospital, Harrow, Middlesex
  - Western General Hospital, Edinburgh, Scotland
  - Taunton And Somerset Hospital, Taunton, Somerset
  - The Institute Of Cancer Research - Royal Marsden Hospital, Sutton, Surrey
  - St Lukes Hospital, Bradford, West Yorkshire
  - Clatterbridge Centre For Oncology, Bebington, WIRRAL
  - Aberdeen Royal Infirmary, Aberdeen
  - Institute Of Cancer Studies - University of Birmingham, Birmingham
  - Royal Sussex County Hospital, Brighton
  - Southmead Hospital, Bristol
  - Addenbrookes Hospital, Cambridge
  - St Richard'S Hospital, Chichester
  - Leighton Hospital, Crewe
  - Gartnavel General Hospital, Glasgow
  - Glasgow Royal Infirmary, Glasgow
  - Freeman Hospital, High Heaton
  - St Batholomew'S Hospital, London
  - Royal Free Hospital, London
  - Clinical Research Centre - St Georges Hospital, London
  - Nottingham City Hospital, Nottingham
  - Derriford Hospital, Plymouth
  - Hope Hospital, Salford
  - Royal Hallamshire Hospital, Sheffield
  - Southampton General, Southampton